CLINICAL TRIAL: NCT00641368
Title: R4Power: An Online Resilience Program for Adolescents
Acronym: R4Power
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swarthmore College (Other)
Responsible Party: Jane E. Gillham, Ph.D., Swarthmore College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-08-003
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Depression; Anxiety
Keywords: Adolescent; Child; Computer; Depression; Resilience
MeSH Terms: conditions — Depression; Anxiety Disorders

ARMS (2):
- 1 (Experimental): R4Power Program
  Interventions: Behavioral: R4Power Program
- 2 (Other): Waitlist Control
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: R4Power Program — In the 10-lesson online R4Power Program, adolescents will learn cognitive skills (link between thoughts, feelings, and behaviors; thinking traps; challenging negative beliefs) and problem-solving skills (assertiveness; relaxation and distraction; overcoming procrastination; decision-making) in order to cope with stressful situations.
  Other Names: R4Power1
  Arms: 1
Other: Waitlist Control — Adolescents in the waitlist control group will complete the R4Power program during the second year of the study.
  Other Names: R4Power2
  Arms: 2

SUMMARY:
The study will evaluate the R4Power program, an online intervention designed to teach adolescents coping and problem-solving skills.

DETAILED DESCRIPTION:
This study examines the feasibility of a 10-lesson web-based intervention, the R4Power program, and its effectiveness in preventing symptoms of depression and anxiety. The R4Power Program teaches cognitive and problem-solving skills covered in classroom based interventions, including the Penn Resiliency Program, that have been found to reduce or prevent symptoms of depression in children and adolescents. This study examines whether adolescents can benefit from learning these skills through a computer (rather than classroom) intervention.

Adolescents in grades 6 through 8 who participate in this study will be assigned to one of two conditions: an intervention group that will complete the R4Power program during the first year (R4Power1), or a waitlist control group that will complete the R4Power program the following year (R4Power2). Students will complete the 10-lesson program over the course of twelve weeks. They will learn and practice cognitive skills (recognizing the link between their thoughts and feelings, identifying thinking traps, challenging their negative beliefs) and problem-solving skills (assertiveness, relaxation and distraction, overcoming procrastination, and decision making). Adolescents who participate in this study will be followed for one year, and their coping responses and symptoms of depression and anxiety will be assessed at four points: at the beginning of the study (baseline) and at follow-up assessments approximately 4, 12 and 16 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* 6th-8th grade students attending participating school OR adolescents aged 11-15 living in greater Philadelphia area
* Access to high speed internet connection (at home, school, or another location)

Exclusion Criteria:

* Below 6th grade reading level, as reported by parents

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Adolescents' coping strategies by self-report | Measured at baseline and follow-ups approximately 4, 12, and 16 months after baseline
Adolescents' depressive symptoms by self-report | Measured at baseline and follow-ups approximately 4, 12, and 16 months after baseline

SECONDARY OUTCOMES:
Adolescents' symptoms of anxiety by self-report | Measured at baseline and follow-ups approximately 4, 12, and 16 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jane E. Gillham, Ph.D., Principal Investigator — Swarthmore College
Locations (1):
- Swarthmore College, Swarthmore, Pennsylvania, United States